CLINICAL TRIAL: NCT03115073
Title: A Phase IIa Randomized, Active-controlled, Double-blind, Dose-escalation Study in Patients With Vulvovaginal Candidiasis to Evaluate Dose Response Relationship of Clinical Efficacy, Safety and Tolerability of Topically Administered ProF-001
Brief Title: ProF-001_Phase IIa
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: ProFem GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ProF-001_Phase IIa
Record Dates: First submitted 2017-03-13; First posted 2017-04-14 (Actual); Last update posted 2019-03-14 (Actual); Status verified 2017-09

CONDITIONS: Vulvovaginal Candidiasis (VVC)
Keywords: Vulvovaginal candidiasis; Candiplus; Clotrimazole; Safety; Tolerability; Clinical efficacy
MeSH Terms: conditions — Candidiasis, Vulvovaginal | interventions — Clotrimazole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- 0,2% Candiplus (Experimental): Candiplus® 0.2%
  Interventions: Drug: Candiplus
- 0,3% Candiplus (Experimental): Candiplus® 0.3%
  Interventions: Drug: Candiplus
- 0,4% Candiplus (Experimental): Candiplus® 0.4%
  Interventions: Drug: Candiplus
- Clotri mono (Active Comparator): Clotrimazole mono
  Interventions: Drug: Clotrimazole

INTERVENTIONS:
Drug: Candiplus — Administration of Candiplus
  Arms: 0,2% Candiplus; 0,3% Candiplus; 0,4% Candiplus
Drug: Clotrimazole — Administration of Clotrimazole
  Arms: Clotri mono

SUMMARY:
This is a multi-center, randomized, prospective, active-controlled, double-blind, dose-escalation study comparing dose response of clinical efficacy, safety, local tolerability of three different doses of ProF-001/Candiplus® (Candiplus® 0.2%, Candiplus® with 0.3%, Candiplus® with 0.4%) to 1% clotrimazole vaginal cream.

Patients with acute episode of vulvovaginal candidiasis (VVC) will be randomized to receive a daily dose of either 5 ml (intravaginal) of Candiplus® at three different doses for the first 3 days and 2.5 ml for the remaining 3 days or 5 ml (intravaginal) application of 1% clotrimazole cream over the first 3 days and 2.5 ml for the remaining 3 days according to the following scheme (with each application 2 cm of cream will be applied to the vulvar region):

Cohort 1: Candiplus® 0.2% versus clotrimazole mono Cohort 2: Candiplus® 0.3% versus clotrimazole mono Cohort 3: Candiplus® 0.4% versus clotrimazole mono Randomization into the cohorts will occur consecutively from the lowest dose to the highest dose, i.e. patients will be randomized first in cohort 1 and finally in cohort 3.

The proposed study is - after a pilot study to assess critical pharmacokinetic data - the second study within a clinical trial program with the objective to develop a new combination therapy for the treatment of vulvovaginal candidiasis.

The new combination consists of two registered drug substances.

ELIGIBILITY:
Inclusion Criteria:

* Premenopausal female patients ≥ 18 years old
* Patients suffering from an acute episode of vulvovaginal candidiasis, characterized by:

  * Positive vaginal smear (native, KOH) for budding yeasts and/or fungal (pseudo-) hyphae, normal or intermediate flora (G I and G II)
  * Positive clinical symptoms (itching, burning, irritation, edema, erythema, excoriations), with a subjective symptom score of at least 3 (0=absent, 1=mild, 2=moderate, and 3=severe), with score being at least moderate for at least 1 subjective symptom and itching being present, and a total sign and symptom score of at least 4
* Readiness for sexual abstinence from start of treatment until test of cure (TOC) - visit
* Sufficient knowledge of German language to understand trial instructions and rating scales, and ability to comply with treatment
* Written informed consent prior to enrolment

Exclusion Criteria:

* Known hypersensitivity to any ingredient of the investigational medicinal product
* Pregnancy or breast feeding at time of screening
* Menstrual bleeding (spotting is not an exclusion criterion) during the first three days of treatment
* Acute cystitis
* Patients with clinical signs of other infectious causes of vulvovaginitis: bacterial vaginosis (GIII), trichomonas vaginalis, herpes simplex genitalis
* Treatment with antimycotics (systemic or vaginal) within 7 days of randomization
* Chronic use of non-steroidal anti-inflammatory drugs (NSAIDs)
* Patients with other clinical gynecological abnormalities, such as infections of the upper urogenital tract (pelvic inflammatory disease, adnexitis)
* Subjects with another vaginal or vulvar condition that would confound the interpretation of clinical response (e.g. Lichen sclerosus, neuropathic pain)
* Subjects who will be under treatment or surgery for gynecological pathologies during the study period, i.e, cervical intraepithelial neoplasia, cervical carcinoma, other neoplasms
* Known alcohol, drug or medication abuse
* Any clinically relevant concomitant condition that could compromise the objectives of this study and/ or the patient's compliance (eg. known immune deficiency syndrome with clinical relevance at time of screening)
* Participation in another interventional clinical trial within the last 30 days
* Employee at the study site, spouse/partner or relative of any study staff (e.g., investigator, sub-investigators, or study nurse) or relationship to the sponsor

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2017-04-04 (Actual); Primary Completion 2018-07-30 (Actual); Study Completion 2018-07-30 (Actual)

PRIMARY OUTCOMES:
Combined outcome measure of: Symptom relief within the first 60 minutes (after application of investigational product or active control) and clinical cure at day 7 (± 3 days). | within 60 minutes after application and at day 7 (± 3 days) after drug application
  As the primary outcome symptom relief within the first 60 minutes will be documented. A reduction of the subjective symptom score ≥ 2 is expected. Furthermore clinical cure at day 7 will be documented. Clinical cure is defined as absence of signs and symptoms of VVC.

SECONDARY OUTCOMES:
Number of patients with local adverse events and serious adverse events (SAEs) with causal relationship to study medication | overall study period (max. 65 days)
  All local adverse events and serious adverse events with causal relationship to study medication (drug reaction) will be documented in a descriptive manner.
Symptom relief within the first 60 minutes (after application of investigational product or active control, reduction of the subjective symptom score ≥ 2) | within 60 minutes after drug application
  Symptom relief within the first 60 minutes will be documented. A reduction of the subjective symptom score ≥ 2 is expected.
Clinical cure (absence of signs and symptoms of VVC) at the TOC visit (=day 7/ accepted time window ±3days) | day 7 ±3 days after drug application
  Clinical cure at day 7 will be documented. Clinical cure is defined as absence of signs and symptoms of VVC.
Mycological outcome: Vaginal swab culture negative for growth of Candida albicans and/or Candida species at the TOC visit (day 7 / ±3days) | day 7 ±3 days after drug application
  A vaginal swab culture will be taken on day 7 / ±3days. The test result is expected to be negative for growth of Candida albicans and/or Candida species.visit (day 7 / ±3days)
Responder outcome: absence of signs and symptoms plus vaginal swab culture negative for growth of Candida albicans and/or Candida species at the TOC visit (day 7 / ±3days) | day 7 ±3 days after drug application
  Presence or absence of signs and symptoms will be documented. Vaginal swab culture is expected to be negative for growth of Candida albicans and/or Candida species at the TOC visit.
Time to improvement of symptoms after first intervention | overall study period (max. 65 days)
  The time to improvement of symptoms after the first intervention will be documented.
Time to termination of clinical symptoms | overall study period (max. 65 days)
  The time to termination of clinical symptoms will be documented.
Clinical relapse of VVC during follow-up period | follow-up period (from day 8 to day 60)
  Every clinical relapse of VVC during the follow-up period will be documented.

CONTACTS AND LOCATIONS:
Overall Officials: Herbert Kiss, Ao.Univ.Prof.Dr., Principal Investigator — Medical University of Vienna
Locations (3):
- Austria (3):
  - Medical University Innsbruck, Innsbruck
  - Bezirkskrankenhaus Schwaz, Schwaz
  - Medical University Vienna, Vienna

REFERENCES:
- [Background] Achkar JM, Fries BC. Candida infections of the genitourinary tract. Clin Microbiol Rev. 2010 Apr;23(2):253-73. doi: 10.1128/CMR.00076-09. PMID 20375352
- [Background] Alem MA, Douglas LJ. Prostaglandin production during growth of Candida albicans biofilms. J Med Microbiol. 2005 Nov;54(Pt 11):1001-1005. doi: 10.1099/jmm.0.46172-0. PMID 16192429
- [Background] Donders G, Bellen G, Byttebier G, Verguts L, Hinoul P, Walckiers R, Stalpaert M, Vereecken A, Van Eldere J. Individualized decreasing-dose maintenance fluconazole regimen for recurrent vulvovaginal candidiasis (ReCiDiF trial). Am J Obstet Gynecol. 2008 Dec;199(6):613.e1-9. doi: 10.1016/j.ajog.2008.06.029. Epub 2008 Oct 30. PMID 18976735
- [Background] Dovnik A, Golle A, Novak D, Arko D, Takac I. Treatment of vulvovaginal candidiasis: a review of the literature. Acta Dermatovenerol Alp Pannonica Adriat. 2015;24(1):5-7. doi: 10.15570/actaapa.2015.2. PMID 25770305
- [Background] Cannom RR, French SW, Johnston D, Edwards JE Jr, Filler SG. Candida albicans stimulates local expression of leukocyte adhesion molecules and cytokines in vivo. J Infect Dis. 2002 Aug 1;186(3):389-96. doi: 10.1086/341660. Epub 2002 Jul 11. PMID 12134235
- [Background] Filler SG, Pfunder AS, Spellberg BJ, Spellberg JP, Edwards JE Jr. Candida albicans stimulates cytokine production and leukocyte adhesion molecule expression by endothelial cells. Infect Immun. 1996 Jul;64(7):2609-17. doi: 10.1128/iai.64.7.2609-2617.1996. PMID 8698486
- [Background] Gale CA, Bendel CM, McClellan M, Hauser M, Becker JM, Berman J, Hostetter MK. Linkage of adhesion, filamentous growth, and virulence in Candida albicans to a single gene, INT1. Science. 1998 Feb 27;279(5355):1355-8. doi: 10.1126/science.279.5355.1355. PMID 9478896
- [Background] Haynes K. Virulence in Candida species. Trends Microbiol. 2001 Dec;9(12):591-6. doi: 10.1016/s0966-842x(01)02237-5. PMID 11728872
- [Background] King RD, Lee JC, Morris AL. Adherence of Candida albicans and other Candida species to mucosal epithelial cells. Infect Immun. 1980 Feb;27(2):667-74. doi: 10.1128/iai.27.2.667-674.1980. PMID 6991423
- [Background] Klotz SA. Fungal adherence to the vascular compartment: a critical step in the pathogenesis of disseminated candidiasis. Clin Infect Dis. 1992 Jan;14(1):340-7. doi: 10.1093/clinids/14.1.340. PMID 1571448
- [Background] Kolachala VL, Bajaj R, Wang L, Yan Y, Ritzenthaler JD, Gewirtz AT, Roman J, Merlin D, Sitaraman SV. Epithelial-derived fibronectin expression, signaling, and function in intestinal inflammation. J Biol Chem. 2007 Nov 9;282(45):32965-73. doi: 10.1074/jbc.M704388200. Epub 2007 Sep 13. PMID 17855340
- [Background] Mathe L, Van Dijck P. Recent insights into Candida albicans biofilm resistance mechanisms. Curr Genet. 2013 Nov;59(4):251-64. doi: 10.1007/s00294-013-0400-3. Epub 2013 Aug 25. PMID 23974350
- [Background] Mendling W, Krauss C, Fladung B. A clinical multicenter study comparing efficacy and tolerability of topical combination therapy with clotrimazole (Canesten, two formats) with oral single dose fluconazole (Diflucan) in vulvovaginal mycoses. Mycoses. 2004 Apr;47(3-4):136-42. doi: 10.1111/j.1439-0507.2004.00970.x. PMID 15078430
- [Background] Muzny CA, Schwebke JR. Biofilms: An Underappreciated Mechanism of Treatment Failure and Recurrence in Vaginal Infections. Clin Infect Dis. 2015 Aug 15;61(4):601-6. doi: 10.1093/cid/civ353. Epub 2015 May 1. PMID 25935553
- [Background] Naglik J, Albrecht A, Bader O, Hube B. Candida albicans proteinases and host/pathogen interactions. Cell Microbiol. 2004 Oct;6(10):915-26. doi: 10.1111/j.1462-5822.2004.00439.x. PMID 15339267
- [Background] Noverr MC, Phare SM, Toews GB, Coffey MJ, Huffnagle GB. Pathogenic yeasts Cryptococcus neoformans and Candida albicans produce immunomodulatory prostaglandins. Infect Immun. 2001 May;69(5):2957-63. doi: 10.1128/IAI.69.5.2957-2963.2001. PMID 11292712
- [Background] Noverr MC, Huffnagle GB. Regulation of Candida albicans morphogenesis by fatty acid metabolites. Infect Immun. 2004 Nov;72(11):6206-10. doi: 10.1128/IAI.72.11.6206-6210.2004. PMID 15501745
- [Background] Nugent RP, Krohn MA, Hillier SL. Reliability of diagnosing bacterial vaginosis is improved by a standardized method of gram stain interpretation. J Clin Microbiol. 1991 Feb;29(2):297-301. doi: 10.1128/jcm.29.2.297-301.1991. PMID 1706728
- [Background] Ray WA, Varas-Lorenzo C, Chung CP, Castellsague J, Murray KT, Stein CM, Daugherty JR, Arbogast PG, Garcia-Rodriguez LA. Cardiovascular risks of nonsteroidal antiinflammatory drugs in patients after hospitalization for serious coronary heart disease. Circ Cardiovasc Qual Outcomes. 2009 May;2(3):155-63. doi: 10.1161/CIRCOUTCOMES.108.805689. Epub 2009 May 5. PMID 20031832
- [Background] Schaller M, Mailhammer R, Korting HC. Cytokine expression induced by Candida albicans in a model of cutaneous candidosis based on reconstituted human epidermis. J Med Microbiol. 2002 Aug;51(8):672-676. doi: 10.1099/0022-1317-51-8-672. PMID 12171298
- [Background] Schaller M, Mailhammer R, Grassl G, Sander CA, Hube B, Korting HC. Infection of human oral epithelia with Candida species induces cytokine expression correlated to the degree of virulence. J Invest Dermatol. 2002 Apr;118(4):652-7. doi: 10.1046/j.1523-1747.2002.01699.x. PMID 11918712
- [Background] Sobel JD, Schmitt C, Stein G, Mummaw N, Christensen S, Meriwether C. Initial management of recurrent vulvovaginal candidiasis with oral ketoconazole and topical clotrimazole. J Reprod Med. 1994 Jul;39(7):517-20. PMID 7966041
- [Background] Sobel JD, Kapernick PS, Zervos M, Reed BD, Hooton T, Soper D, Nyirjesy P, Heine MW, Willems J, Panzer H, Wittes H. Treatment of complicated Candida vaginitis: comparison of single and sequential doses of fluconazole. Am J Obstet Gynecol. 2001 Aug;185(2):363-9. doi: 10.1067/mob.2001.115116. PMID 11518893
- [Background] Theraud M, Bedouin Y, Guiguen C, Gangneux JP. Efficacy of antiseptics and disinfectants on clinical and environmental yeast isolates in planktonic and biofilm conditions. J Med Microbiol. 2004 Oct;53(Pt 10):1013-1018. doi: 10.1099/jmm.0.05474-0. PMID 15358824
- [Background] Thompson DS, Carlisle PL, Kadosh D. Coevolution of morphology and virulence in Candida species. Eukaryot Cell. 2011 Sep;10(9):1173-82. doi: 10.1128/EC.05085-11. Epub 2011 Jul 15. PMID 21764907
- See also: Lisa A. Bero, February 15, 2005, Expert Committee on Selection and Use of Essential Medicines, Review of Application of Clotrimazole for topical or intravaginal use in vulvovaginal candidiasis. — http://archives.who.int/eml/expcom/expcom14/clotrimazole/clotrimazole_ECP_review_16feb05.pdf
- See also: FDA draft Guidance for Industry Vulvovaginal Candidiasis -Developing Drugs for Treatment, 2016. — http://www.fda.gov/downloads/Drugs/GuidanceComplianceRegulatoryInformation/Guidances/UCM509411.pdf
- See also: Newcombe, R.G. "Interval estimation for the difference between independent proportions: comparison of eleven methods" Statistics in Medicine 17(1988) pp. 873-890 — https://pdfs.semanticscholar.org/370b/92bc4f61fedfa64e1b50e7a10c7a6dde0a19.pdf
- See also: Santoni G, Gismondi A, Liu JH, et al. Candida albicans expresses a fibronectin receptor antigenically related to a5b1 integrin. Microbiology. 1994 Nov;140 ( Pt 11):2971-9. — http://mic.microbiologyresearch.org/content/journal/micro/10.1099/13500872-140-11-2971
- See also: Voltarol Suppositories 12.5 mg, 25 mg, 50 mg, 100 mg, UK SmPC 2013 — https://www.medicines.org.uk/emc/medicine/1344